CLINICAL TRIAL: NCT05403008
Title: Clinical Performance and Wear Resistance of Highly Translucent Nano Zirconia Reinforced Glass Ionomer Filling Versus Conventional Resin Composite Restorations in Patients With Proximal Carious Teeth. (A One-year Randomized Clinical Trial).
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Weaam Mohamed Abdelfatah Abdelfatah Ammar, Master degree student, Conservative Dentistry Department, Faculty of Dentistry, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Zirconomer Improved
Record Dates: First submitted 2022-02-02; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessors and statistician
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zirconomer improved (Other): a nano zirconia reinforced glass ionomer, which has improved the mechanical, esthetic and handling properties than its previous successor.
  Interventions: Other: Zirconomer improved
- Nano hybird resin composite (Active Comparator): Resin composite (RC) is the gold standard esthetic restoration in proximal cavities due to their high aesthetic properties, increased mechanical durability and enhanced adhesion to tooth structure.
  Interventions: Other: Zirconomer improved

INTERVENTIONS:
Other: Zirconomer improved — Zirconomer improved, is a nano zirconia reinforced glass ionomer, which has improved the mechanical, esthetic and handling properties than its previous successor.

SUMMARY:
This randomized clinical study aims to evaluate the clinical performance and occlusal wear resistance of nano-zirconia reinforced glass ionomer restorations in comparison to Nano-hybrid resin composite in proximal cavities.

DETAILED DESCRIPTION:
Statement of the problem:

The glass ionomer restorations have a wide use in dental community. Proximal restoration is a challenge, due to the high forces present in this area that require more high fracture resistance restoration material which is not obtained in the most of the versions of glass ionomer restorations that are available in dental market.(Safy, 2019)

Rationale for choice of intervention:

Zirconomer improved, is a nano zirconia reinforced glass ionomer, which has improved the mechanical, esthetic and handling properties than its previous successor, zirconomer. Zirconomer is commercialized as a white amalgam as it features mechanical properties similar to amalgam restorations. In this generation also, translucency is improved to be similar to the tooth structure.(Shetty et al, 2017) As Zirconomer improved is reinforced material, it is expected that has high wear resistance than the conventional glass ionomer restorations. (Hesse et al., 2018)

ELIGIBILITY:
Inclusion Criteria:

* Age group 18-55
* Presence of occluding tooth.
* Good oral hygiene

Exclusion Criteria:

* Poor periodontal status
* Adverse medical history.
* Potential behavioral problems

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2022-06 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Postoperative Hypersensitivity Secondary caries
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Secondary caries and measured by Modified United States Public Health Service Criteria (USPHS)
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Gross fracture and measured by Modified United States Public Health Service Criteria (USPHS)
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Color match and measured by Modified United States Public Health Service Criteria (USPHS)
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Cavo-surface marginal discoloration and measured by Modified United States Public Health Service Criteria (USPHS)
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Marginal integrity and measured by Modified United States Public Health Service Criteria (USPHS)
Clinical performance | Change from the baseline at 6 months and at 12 months.
  Proximal contact and measured by Modified United States Public Health Service Criteria (USPHS)

SECONDARY OUTCOMES:
Wear resistance evaluation | Change from the baseline at 6 months and at 12 months.
  "Wear measurements Measured by using WSxM software.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed El-Hoshy, Professor, Study Director — Cairo University